CLINICAL TRIAL: NCT00086736
Title: A Randomized, Placebo-Controlled Phase IIb Clinical Trial of 2-Difluoromethylornithine (DFMO) Versus Bicalutamide (CASODEX) Alone and in Combination in Patients With Prostate Cancer in the Period Prior to Radical Prostatectomy or Brachytherapy: Modulation of Tissue and Molecular Biomarkers in Human Prostate Tissue Serum
Brief Title: Neoadjuvant Eflornithine and Bicalutamide Compared With Eflornithine Alone, Bicalutamide Alone, and No Neoadjuvant Therapy in Treating Patients With Localized Prostate Cancer Undergoing Brachytherapy or Radical Prostatectomy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CDR0000353198; UAB-9921; UAB-F990728039
Record Dates: First submitted 2004-07-08; First posted 2004-07-12 (Estimated); Last update posted 2013-11-19 (Estimated); Status verified 2013-07

CONDITIONS: Prostate Cancer
Keywords: stage I prostate cancer; stage IIB prostate cancer; stage IIA prostate cancer; stage III prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — bicalutamide; Eflornithine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Arm I (Experimental): Patients receive oral eflornithine and oral bicalutamide once daily for 28 days in the absence of unacceptable toxicity. Patients then undergo either prostatectomy or brachytherapy, as determined by the patient, on day 29.
  Interventions: Drug: bicalutamide; Drug: eflornithine
- Arm II (Experimental): Patients receive oral eflornithine and oral bicalutamide placebo once daily for 28 days in the absence of unacceptable toxicity. Patients then undergo either prostatectomy or brachytherapy, as determined by the patient, on day 29.
  Interventions: Drug: eflornithine; Drug: oral bicalutamide placebo
- Arm III (Experimental): Patients receive oral eflornithine placebo and oral bicalutamide once daily for 28 days in the absence of unacceptable toxicity. Patients then undergo either prostatectomy or brachytherapy, as determined by the patient, on day 29.
  Interventions: Drug: bicalutamide; Drug: oral eflornithine placebo
- Arm IV (Experimental): Patients receive oral eflornithine placebo and oral bicalutamide placebo once daily for 28 days in the absence of unacceptable toxicity. Patients then undergo either prostatectomy or brachytherapy, as determined by the patient, on day 29.
  Interventions: Drug: oral eflornithine placebo; Drug: oral bicalutamide placebo

INTERVENTIONS:
Drug: bicalutamide
  Arms: Arm I; Arm III
Drug: eflornithine
  Arms: Arm I; Arm II
Drug: oral eflornithine placebo
  Arms: Arm III; Arm IV
Drug: oral bicalutamide placebo
  Arms: Arm II; Arm IV

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as eflornithine, work in different ways to stop tumor cells from dividing so they stop growing or die. Androgens can stimulate the growth of prostate cancer cells. Drugs used in hormone therapy, such as bicalutamide, may fight prostate cancer by stopping the adrenal glands from producing androgens. Combining eflornithine with bicalutamide may kill more tumor cells.

PURPOSE: Randomized phase II trial to compare the effectiveness of neoadjuvant eflornithine and bicalutamide with that of eflornithine alone, bicalutamide alone, and no neoadjuvant therapy in treating patients who are undergoing brachytherapy or radical prostatectomy for localized prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare levels of polyamine spermine, polyamine putrescine, and spermidine in patients with localized prostate cancer undergoing brachytherapy or radical prostatectomy and treated with neoadjuvant eflornithine and bicalutamide vs eflornithine alone vs bicalutamide alone vs no neoadjuvant therapy.
* Compare the expression of surrogate biomarkers (i.e., serum prostate-specific antigen, tissue levels of proliferating cell nuclear antigen, Ki67, and TGF-alpha, apoptosis assays [ICH-PARP and TUNEL], and cytomorphometric indices) in patients treated with these regimens.
* Compare the toxicity of these regimens in these patients.

OUTLINE: This is a randomized, double-blind, placebo-controlled study. Patients are stratified according to Gleason score (< 7 vs ≥ 7). Patients are randomized to 1 of 4 treatment arms.

* Arm I: Patients receive oral eflornithine and oral bicalutamide once daily.
* Arm II: Patients receive oral eflornithine and oral bicalutamide placebo once daily.
* Arm III: Patients receive oral eflornithine placebo and oral bicalutamide once daily.
* Arm IV: Patients receive oral eflornithine placebo and oral bicalutamide placebo once daily.

In all arms, treatment continues for 28 days in the absence of unacceptable toxicity. Patients then undergo either prostatectomy or brachytherapy, as determined by the patient, on day 29.

Patients are followed at 4 weeks.

PROJECTED ACCRUAL: A total of 44 patients (11 per treatment arm) will be accrued for this study within 11 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed prostate cancer

  * Localized disease
* Paraffin blocks from diagnostic biopsies available
* Planning to undergo brachytherapy or prostatectomy

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-3

Life expectancy

* Not specified

Hematopoietic

* Hemoglobin ≥ 10.0 g/dL
* WBC ≥ 3,500/mm^3
* Platelet count ≥ 125,000/mm^3

Hepatic

* Bilirubin ≤ 2.0 mg/dL
* SGOT and SGPT ≤ 2 times normal
* No history of liver disease (e.g., hepatitis, cirrhosis, or jaundice)

Renal

* Creatinine ≤ 2.0 mg/dL

Cardiovascular

* No symptomatic coronary artery disease
* No uncontrolled hypertension
* No acute myocardial infarction within the past year

Other

* Fertile patients must use effective contraception
* No more than 10 decibels baseline hearing loss at any frequency by full bilateral audiometry within the past month
* No hypersensitivity to eflornithine or bicalutamide
* No other prior or active malignancy except nonmelanoma skin cancer or other cancer curatively treated at least 5 years ago with no evidence of recurrent or residual disease
* No concurrent acute or chronic medical or psychiatric condition that would preclude study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No concurrent immunotherapy

Chemotherapy

* No other concurrent chemotherapy

Endocrine therapy

* More than 1 year since prior antiandrogen, luteinizing hormone-releasing hormone (LHRH) agonist, bicalutamide, finasteride, or diethylstilbestrol
* No other concurrent antiandrogen, LHRH agonist, finasteride, or diethylstilbestrol

Radiotherapy

* See Disease Characteristics
* No other concurrent radiotherapy

Surgery

* See Disease Characteristics

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2001-11; Primary Completion 2003-11 (Actual); Study Completion 2003-11 (Actual)

PRIMARY OUTCOMES:
Mean difference in levels of Polyamine spermine, polyamine putrescine, and spermidine between subjects in each of the 4 groups | 4 weeks after surgical intervention

CONTACTS AND LOCATIONS:
Overall Officials: Donald A. Urban, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham Comprehensive Cancer Center, Birmingham, Alabama, United States